CLINICAL TRIAL: NCT05280990
Title: HepaRAS Trial: Changes in Hepatectomy Risk Assessment When Incorporating Mebrofenin HIDA for Functional Evaluation of the Liver Remnant: A Pilot Study
Brief Title: HepaRAS Trial: Changes in Hepatectomy Risk Assessment When Using Mebrofenin HIDA
Acronym: HepaRAS
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Technical requirements not met.
Sponsor: Boris Gala Lopez (Other)
Collaborators: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Sponsor-Investigator, Boris Gala Lopez, Assistant Professor, Nova Scotia Health Authority
Organization: Nova Scotia Health Authority (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 45465
Record Dates: First submitted 2022-03-06; First posted 2022-03-15 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Liver Failure as A Complication of Care; 30-day Mortality

STUDY DESIGN:
Intervention Model Description: Hypothesis: Using Future Liver Remnant Function (FLRF) through 99mTc-mebrofenin hepatobiliary scintigraphy (mHBS) to select patients for major hepatectomy will reduce the rate of Post-hepatectomy liver failure (PHLF), compared to our standard-of-care Future Liver Remnant Volume (FLRV) calculations for patient selection.
  Methods: This is a prospective pilot study designed to evaluate feasibility and safety in the Canadian settings and will include patients undergoing major liver resection at the Queen Elizabeth II Health Sciences Centre (QEII) in Halifax, Canada, and at McGill University Health Centre in Montreal, Canada (McGill). Recruited patients, irrespective of their underlying liver quality will be randomly assigned via block randomization to have either preoperative FLRV assessment by CT/MRI volumetry or preoperative FLRF risk assessment via mHBS.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Future Liver Remnant Function (FLRF) (Experimental): Preoperative FLRF risk assessment via 99mTc-mebrofenin hepatobiliary scintigraphy (mHBS)
  Interventions: Diagnostic Test: mHBS
- Future Liver Remnant Volume (FLRV) (Active Comparator): Preoperative FLRV assessment by CT/MRI volumetry
  Interventions: Diagnostic Test: CT/MRI volumetry

INTERVENTIONS:
Diagnostic Test: mHBS — Preoperative FLRF assessment using 99mTc-mebrofenin hepatobiliary scintigraphy (mHBS).
  Arms: Future Liver Remnant Function (FLRF)
Diagnostic Test: CT/MRI volumetry — Preoperative FLRF assessment using CT/MRI volumetry
  Arms: Future Liver Remnant Volume (FLRV)

SUMMARY:
Surgical procedures to remove a significant portion of the liver are used to treat various diseases including cancer. They have demonstrated to be the most effective treatment for selected patients. These procedures rely on the fascinating ability of the liver to grow back, allowing surgeons to remove of up to 70% of the organ in a safe manner. However, there are instances where severe complications and death occur due to the inability of the residual liver to perform all functions. It is estimated that up to 32% of patients undergoing this type of surgery will experience such complications. To prevent this, physicians calculate the total liver volume before surgery using radiology and estimate how much liver will remain after surgery. Only when the liver remnant is 30% or higher, the procedure is deemed safe.

One of the main limitations of this strategy is that the estimated percentage of the liver remnant does not entirely reflect a proportional function. To overcome this limitation and avoid serious complications, a more precise assessment is required. Recently, a new scan was introduced using mebrofenin, which is metabolized in the liver and can be traced in a particular region of the organ using computer software. As a result, clinicians can know with certainty, the percentual function of a portion of the liver, and if that portion will be sufficient to avoid complications and death after a major liver operation.

This project proposes incorporating this technology for preoperative evaluation against our traditional assessment using just volume calculations. Participants will be randomly assigned to the traditional volume calculation or the new scan with mebrofenin, and investigators will compare how well both methods are able to predict complications and death after surgery. Researchers are particularly interested in demonstrating if major complications and death after surgery are less using the new mebrofenin scan.

Our study evaluating the introduction of a new and relatively harmful technique will help to better identify those patients with high risk for complications and death after a major surgical procedure on the liver. This will help in better selecting future patients and will allow for a more precise discussion during initial evaluation.

DETAILED DESCRIPTION:
Surgical procedures to remove a significant portion of the liver are used to treat various diseases, including cancer. They have been demonstrated to be the most effective treatment for selected patients. These procedures rely on the fascinating ability of the liver to grow back, allowing surgeons to remove up to 70% of the organ in a safe manner. However, there are instances where severe complications and death occur due to the inability of the residual liver to perform all functions. It is estimated that up to 32% of patients undergoing this type of surgery will experience such complications. To prevent this, physicians use radiology to calculate the total liver volume before surgery and estimate how much liver will remain after surgery. The procedure is deemed safe only when the liver remnant is 30% or higher.

One of the main limitations of this strategy is that the estimated percentage of the liver remnant does not entirely reflect a proportional function. A more precise assessment is required to overcome this limitation and avoid serious complications. Recently, a new scan was introduced using computer software using mebrofenin, which is metabolized in the liver and can be traced in a particular organ region. As a result, clinicians can know with certainty the percentual function of a portion of the liver and if that portion will be sufficient to avoid complications and death after a major liver operation.

This project proposes incorporating this technology for preoperative evaluation against our traditional assessment using just volume calculations. Participants will be randomly assigned to the traditional volume calculation or the new scan with mebrofenin, and investigators will compare how well both methods are able to predict complications and death after surgery. Researchers are particularly interested in demonstrating if major complications and death after surgery are less common using the new mebrofenin scan.

Our study evaluating the introduction of a new and relatively harmful technique will help to better identify those patients with a high risk for complications and death after a major surgical procedure on the liver. This will help better select future patients and allow for a more precise discussion during the initial evaluation.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients who are being considered for major hepatectomy at the QEII and McGill for malignant or benign disease.
* Both open and laparoscopic approaches will be accepted in the study.
* Patients with underlying liver cirrhosis or receiving additional ablation therapies will not be excluded.

Exclusion Criteria:

* Patients younger than 18 years-old.
* Pregnant patients.
* Hepatectomy is associated with another major non-liver procedure.
* Patients not qualifying for a major hepatectomy following preoperative assessment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-01-15 (Estimated); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-07-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants with post-hepatectomy liver failure (PHLF) | 30 days
  Incidence of post-hepatectomy liver failure (PHLF)

SECONDARY OUTCOMES:
Number of participants with the 50-50 criteria | 5 days
  Prothrombin time <50% of normal and serum bilirubin >50 µmol/L on POD 5, which is an early predictor of more than 50% mortality rate after hepatectomy.
Number of participants with major postoperative complications as per Clavien-Dindo classification | 30 days
  Occurrence of major postoperative complications as per Clavien-Dindo classification
Hospital length of stay | 30 days
  Hospital length of stay
30-day mortality | 30 days
  30-day mortality

CONTACTS AND LOCATIONS:
Overall Officials: Boris Gala-Lopez, MD, MSC, PhD, Principal Investigator — Queen Elizabeth II Health Sciences Centre. Dalhousie University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Guglielmi A, Ruzzenente A, Conci S, Valdegamberi A, Iacono C. How much remnant is enough in liver resection? Dig Surg. 2012;29(1):6-17. doi: 10.1159/000335713. Epub 2012 Mar 15. PMID 22441614
- [Background] Gupta M, Choudhury PS, Singh S, Hazarika D. Liver Functional Volumetry by Tc-99m Mebrofenin Hepatobiliary Scintigraphy before Major Liver Resection: A Game Changer. Indian J Nucl Med. 2018 Oct-Dec;33(4):277-283. doi: 10.4103/ijnm.IJNM_72_18. PMID 30386047
- [Background] de Graaf W, van Lienden KP, Dinant S, Roelofs JJ, Busch OR, Gouma DJ, Bennink RJ, van Gulik TM. Assessment of future remnant liver function using hepatobiliary scintigraphy in patients undergoing major liver resection. J Gastrointest Surg. 2010 Feb;14(2):369-78. doi: 10.1007/s11605-009-1085-2. PMID 19937195
- [Background] Bennink RJ, Dinant S, Erdogan D, Heijnen BH, Straatsburg IH, van Vliet AK, van Gulik TM. Preoperative assessment of postoperative remnant liver function using hepatobiliary scintigraphy. J Nucl Med. 2004 Jun;45(6):965-71. PMID 15181131